CLINICAL TRIAL: NCT01611480
Title: Efficacy and Safety of a New Topical Formulation With Imiquimod (Limtop) Applied 1, 3 or 7 Times Weekly During 2 x 2 Weeks Treatment for Actinic Keratosis on the Head
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: LIMTOP-I
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

INTERVENTIONS:
Drug: Imiquimod (topical use)

SUMMARY:
The aim is to evaluate efficacy and safety of three different dosing regimens of Limtop in a study involving 96 patients with actinic keratosis on the head or face.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form (ICF) signed and dated by the patient prior to any study-related activity
2. Male or female patients aged 18 or older
3. Have a total of 5-20 clinically confirmed, palpable or visible (grade I or II according to modified Olsen score) nonhyperkeratotic, nonhypertrophic AK lesions located within a contiguous 25 - 100 cm² area on the balding scalp or face
4. Any skin type or race, providing the skin pigmentation will allow discernment of erythema
5. Willingness to actively participate in the study and to comply with the study procedures as defined in the study protocol
6. High probability of a good compliance and orderly completion of the study
7. Negative urine pregnancy test (in female subjects with childbearing potential)

   -

Exclusion Criteria:

1. Evidence of clinically significant, unstable cardiovascular or immunosuppressive, hematologic, hepatic, neurologic, renal, endocrine, collagen-vascular, or gastrointestinal abnormalities or disease
2. Diagnosed autoimmune diseases and anaemia
3. Any dermatological disease and or condition in the treatment or surrounding area that may be exacerbated by treatment with imiquimod or cause difficulty with examination (e.g. rosacea, psoriasis, atopic dermatitis, eczema)
4. Any significant findings (e.g. tattoos) in the potential application site area that may impair examination of treatment or surrounding area
5. Confirmed squamous cell or basal cell carcinoma anywhere on the head in the past 3 months
6. Share a household where there is a person participating in a concurrent clinical study of imiquimod or being treated with imiquimod 5% topical cream
7. Active chemical dependency or alcoholism, as assessed by investigator
8. Patients unwilling to stay out of the sun or wear protective clothing or to take appropriate measures to cover the treatment area during the study
9. Previous treatments with imiquimod for AK in the predetermined treatment area within the past 3 months
10. Treatment with COX-2 inhibitors 14 days prior to randomization
11. Currently using or have used on the treatment area over-the-counter retinol products, corticosteroids, cryosurgery, curettage, 5-fluorouracil, or other topical actinic keratosis treatments 28 days prior to randomization
12. Subjects who experienced an unsuccessful outcome from previous imiquimod therapy.
13. Known allergy or sensitivity to imiquimod or any of the excipients (butyl lactate, isopropyl myristate, propylene glycol, butylated hydroxy anisole) in the IMP
14. Pre-menopausal (last menstruation ≤ 1 year prior to screening) sexually active women who:

    * are pregnant or nursing,
    * are not surgically sterile,
    * are of child bearing potential and not practicing an acceptable method of birth control, or does not plan to continue practicing an acceptable method of birth control throughout the trial (acceptable methods include intrauterine devices (IUD), oral, implantable or injectable contraceptives, diaphragm or cervical cap with intravaginal spermicide, condom with intravaginal spermicide or vasectomised partner)
15. Participation in another clinical trial with an investigational drug or device during the previous 4 weeks before Baseline
16. Receiving systemic cancer chemotherapy, psoralen plus UVA therapy, UVB therapy, laser abrasion, dermabrasion, glycolic acids, or chemical peels 6 months prior to study entry.
17. Currently using or have used systemic steroids 2 months prior to study except inhaled corticosteroids (<1200 microgram/day for beclomethasone, or <600 microgram/day for fluticasone)
18. Known infectious diseases (e.g. HIV, hepatitis)
19. Psychiatric condition that might limit the participation in the study and/or that lead to the assumption that the ability to completely understand the consequences of consent is missing
20. The Patient is institutionalized by virtue of an order issued either by the judicial or the administrative authorities
21. Employee of the study site or of the Sponsor's company
22. Any disease or circumstances on account of which the subject should not participate in the study in the opinion of the investigator -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 5 Locations, Germany, Germany